CLINICAL TRIAL: NCT03551665
Title: Effects of Protective Step Training in People With Multiple Sclerosis
Brief Title: Protective Stepping in People With MS
Acronym: PRO-STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2341-W
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Falls; Posture; Rehabilitation; Cognition; Neuroimaging
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Multiple-baseline, within-subject design
Masking Description: Primary outcomes are objective (i.e. assessed via computer algorithms), thus reducing the need for masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Step training (Experimental): This group will undergo a baseline control period, as well as an intervention period. As such, they will serve as their own control subjects.
  Interventions: Behavioral: Protective step training

INTERVENTIONS:
Behavioral: Protective step training — Participants will undergo 2 weeks of training, in which they will be exposed to repeated slips on a treadmill. This approach is aimed at improving protective steps.

SUMMARY:
Falls are common in Veterans with multiple sclerosis (MS), and current rehabilitation approaches to reduce falls are inadequate. Protective step training (in which a person is exposed to repeated "slips") is a promising tool to reduce falls in older adults. However, whether this approach is effective in people with MS is unknown. Investigating the effect of promising therapies, such as protective step training, will enhance our ability to treat Veterans with MS who are at risk for falls. Therefore, we will assess whether people with MS improve postural control and reduce falls through protective step training. we will also determine whether cognitive ability or brain structure can predict who will improve most. These data will inform clinical treatment strategies in people with MS at risk for falls.

DETAILED DESCRIPTION:
Current rehabilitation strategies to prevent falls in people with MS are inadequate. Protective step training is a novel and promising treatment in which people are exposed to repeated slips. This training aims to improve automatic postural control including quick, protective steps, which are a critical aspect of fall avoidance, and are delayed in people with MS. This therapy has been shown to prevent falls in healthy older adults. However, the effectiveness of perturbation training in Veterans with MS is unknown. Identifying effective methods of fall prevention in people with MS, such as perturbation training, can lead to fewer falls in this population.

People with MS often exhibit considerable variability in their "responsiveness" to rehabilitation. Said differently, improvement in performance through training is variable across individuals. The ability to predict responsiveness to treatment would be extremely beneficial for clinicians; improving the efficiency by which they provide care. Recent work suggests cognitive ability and structural brain connectivity may predict responsiveness to motor rehabilitation. However, the degree to which these characteristics predict responsiveness in people with MS is currently unknown.

Therefore, the overall goals of this project are to understand 1) whether people with MS can improve postural control and reduce falls through perturbation training, and 2) whether the investigators can predict (via cognitive testing and neuroimaging), who will benefit most from treatment. The investigators will achieve these goals through three specific aims. Aim 1: identify whether people with MS can improve protective stepping, a critical skill for fall prevention, through 2 weeks of protective step training. Aim 2: determine if cognitive capacity predicts postural improvement through training in people with MS. Aim 3: determine if brain structural connectivity predicts postural improvements through training. The imaging data collected will also allow the investigators to investigate whether MS-related changes in brain connectivity contributes to postural response dysfunction.

The efficacy of perturbation training in people with MS (Aim 1) will be studied by measuring protective stepping performance before and after a 2-week perturbation training protocol. In addition, the investigators will gather prospective falls data through a falls calendar over the course of 8 weeks prior to and 8 weeks after the perturbation training to gain preliminary data regarding the effect of this training on falls. To determine which baseline characteristics predict "responsiveness" to training (Aims 2 and 3), the investigators will also assess baseline cognitive capacity and brain structural integrity (via diffusion tensor imaging; DTI). The investigators will determine whether these baseline participant characteristics predict which participants exhibit the most improvement through the course of training.

This project will provide insight into 1) the effectiveness of a promising fall prevention intervention, and 2) the ability to predict which patients will benefit most from the intervention. This knowledge will be an important step toward improving care of people with MS who are at risk for falls.

ELIGIBILITY:
Inclusion Criteria:

* Neurologist diagnosed MS (for MS participants only)
* Ability to Stand for 5 minutes without aid
* Ability to comprehend English
* At risk for falls (determined via questionnaire; for MS participants only)
* EDMUS score <7 (determined by testers)

Exclusion Criteria:

* Any non-MS neurological pathology
* Orthopedic impairments affecting balance
* Previous cardiac events (stroke or heart attack)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Peterson, PhD MS BS, Principal Investigator — Phoenix VA Health Care System, Phoenix, AZ
Locations (1):
- Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be collected at Arizona State University, and thus will be accessible by study-team members at this institution.
Supporting Information: Study Protocol, SAP
Time Frame: Data collected at ASU will be stored indefinitely.
Access Criteria: Only approved study-team members at ASU will have access to IPD. These individuals will be identified and personally trained by the PI on the grant (Dr. Peterson).

RESULTS

PARTICIPANT FLOW:
Groups:
- Step Training (MS Group): This group of people with MS will undergo a baseline control period, as well as an intervention period. As such, they will serve as their own control subjects.
- Step Training (Control Group): This group of people without MS will undergo a baseline control period, as well as an intervention period. As such, they will serve as their own control subjects.
Period: Overall Study
Arm/Group | Step Training (MS Group) | Step Training (Control Group)
Started | 38 | 19
Completed | 27 | 17
Not Completed | 11 | 2
Not completed — Lost to Follow-up | 11 | 2

BASELINE CHARACTERISTICS:
Population: 57 people were originally screened and enrolled (38 MS and 19 control). Of these, 44 completed the baseline testing and are included in further analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Step Training (MS Group) | Step Training (Control Group) | Total
Number analyzed (Participants) | 27 | 17 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years Population: 57 people were originally screened and enrolled (38 MS and 19 control). Of these, 44 completed the baseline testing.
  years | 56.49 (13.97) | 58.31 (19.30) | 57.20 (16.04)
Sex: Female, Male [Count of Participants; unit: Participants] — 57 people were originally screened and enrolled (38 MS and 19 control). Of these, 44 completed the baseline testing and are included in further analyses.
  Participants
    Female | 16 | 11 | 27
    Male | 11 | 6 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants] — 57 people were originally screened and enrolled (38 MS and 19 control). Of these, 44 completed the baseline testing and are included in further analyses.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 0 | 2
    White | 25 | 15 | 40
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 27 | 14 | 41
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Training-related Change in Margin of Stability
Description: Margin of Stability is a measure of stepping effectiveness; characterized as the difference between the extrapolated center of mass and the base of support at the instance of first foot contact. The primary endpoint was the change in Margin of Stability before to after training (i.e. Baseline to Post-test). The units of this measure are in meters. Large values represent better steps. So, positive change scores represent improvement in stepping.
Time Frame: Baseline and Post-test (immediately after the intervention)
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Step Training (MS Group): People with multiple sclerosis
- Step Training (Control Group): People without MS.
Arm/Group | Step Training (MS Group) | Step Training (Control Group)
Number analyzed (Participants) | 27 | 17
meters | 0.0289 (0.0777) | 0.0217 (0.119)
Statistical Analysis 1: Comparison: Step Training (MS Group); These data are the immediate improvements (base 2 - post 1) in the MS group; Test type: Other; p = 0.036, Regression, Linear; Mean Difference (Final Values) = .029, 95% CI 2-sided [.002 to 0.056]

2. Primary Outcome: Symbol Digit Modality Test
Description: The Symbol Digit Modality Test (SDMT) is a cognitive assessment that probes processing speed. The score is the number of symbols and digits that one correctly matches over 90 seconds, and is assessed via paper and pencil. As such, the lower bound is 0, and there is no upper bound. Larger values are better.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- MS Group: People with MS
- Step Training (Control Group): Individuals without multiple sclerosis
Arm/Group | MS Group | Step Training (Control Group)
Number analyzed (Participants) | 27 | 17
Units on a scale | 42.44 (10.33) | 51.88 (8.44)
Statistical Analysis 1: Comparison: MS Group; We correlated cognition (SDMT; above) to the improvement in performance (margin of stability) to to determine whether cognition predicted improvement in stepping outcomes; Test type: Other; p = .92, Spearman Correlation; Spearman's Rho = .019

3. Secondary Outcome: Training-related Changes in Reactive Step Length
Description: Reactive Step Length is the length of the first step after the participant loses their balance. The primary endpoint was the immediate change in performance through training (i.e., initial training period; Base2-Post1). The primary endpoint was the change in Reactive Step Length before to after training (i.e., Baseline to Post-test). The units of this measure are in meters. Large values represent better steps. So, positive change scores represent improvement in stepping.
Time Frame: Baseline and Post-test (immediately after the intervention)
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Step Training (Control Group): People without multiple sclerosis
Arm/Group | Step Training (MS Group) | Step Training (Control Group)
Number analyzed (Participants) | 27 | 17
meters | 0.026 (0.086) | 0.023 (0.063)
Statistical Analysis 1: Comparison: Step Training (MS Group); We assessed the change in reactive step length before (Baseline 2) to immediately after (post 1) training in the MS group; Test type: Other; p = 0.119, Regression, Linear; Mean Difference (Final Values) = 0.026, 95% CI [-0.007 to 0.059]

4. Secondary Outcome: Training-related Change in Reactive Step Latency
Description: Reactive Step Latency is the time between when the balance perturbation occurs to lift-off of the foot. The primary endpoint was the change in performance through training (i.e., Baseline to Post-test). Smaller values represent faster (better) steps. So, negative change scores represent improvement in stepping through training.
Time Frame: Baseline and Post-test (immediately after 2 week intervention)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Step Training (MS Group) | Step Training (Control Group)
Number analyzed (Participants) | 27 | 17
seconds | -0.0414 (0.1047) | 0.0047 (0.0500)
Statistical Analysis 1: Comparison: Step Training (MS Group); We assessed the change in reactive step latency before (Baseline 2) to immediately after (post 1) training in the MS group; Test type: Other; p = 0.012, Regression, Linear; Mean Difference (Final Values) = -0.041, 95% CI [-0.073 to -0.009]

ADVERSE EVENTS:
Time Frame: Across the training period (2 weeks)
Arm/Group | Step Training (MS Group) | Step Training (Control Group)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/17
Other Adverse Events (participants affected / at risk) | 0/27 | 0/17

LIMITATIONS AND CAVEATS:
Technical problems with neuroimaging data analyses have resulted in unreliable or uninterpretable data at this time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT03551665/Prot_SAP_000.pdf